CLINICAL TRIAL: NCT02325856
Title: Effect of Post-dialysis Weight Evaluated With Bioimpedance Spectroscopy on Dialysis Morbidities and Clinical Outcomes in Hemodialysis Patients: A Randomized Controlled Trial
Brief Title: Application of Bioimpedance Spectroscopy in Taiwan Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: An Hsin QingShui Clinic (Other)
Collaborators: Nephrocare AsiaPacific (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ABISAD-3
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Results first posted 2015-08-17 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2015-07

CONDITIONS: Fluid Overload
Keywords: Hemodialysis; Body Composition Monitor
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Active Comparator): Dry weight determined by performing Bioimpedance Spectroscopy (intervention is the performance of this tool)
  Interventions: Device: Bioimpedance Spectroscopy
- Control group (Placebo Comparator): Dry weight determined by clinical symptoms
  Interventions: Behavioral: Clinical judgement

INTERVENTIONS:
Device: Bioimpedance Spectroscopy — Bioimpedance Spectroscopy is a safe tool to evaluate the fluid status in hemodialysis patients.
  Arms: Study group
Behavioral: Clinical judgement
  Arms: Control group

SUMMARY:
A reasonable and simple algorithm was used to guide the dry weight determination with Body Composition Monitor with the principle of Bioimpedance Spectroscopy (BCM-BIS) and analyze the feasibility of this algorithm and evaluate the influence of BCM-BIS-guided fluid management on the incidence of dialysis morbidities and clinical outcomes in maintenance hemodialysis (MHD) patients.

DETAILED DESCRIPTION:
298 MHD patients in 6 hemodialysis centers in Taiwan were enrolled in this randomized controlled study. All the participants were randomized into study group ( dry weight (DW) determined by BCM-BIS) and control group ( dry weight determined by clinical symptoms) with stratification by diabetes mellitus and centers. Body composition monitor based on bioimpedance spectroscopy (BCM-BIS) was performed monthly and concomitant biochemical data and clinical outcomes were collected. Intra-dialysis complications were recorded in every dialysis session. Primary outcome was all-cause hospitalization. Secondary outcomes included 1) complications during DW adjustment 2) intra-dialysis morbidities 3) hypertension 4) mortality 5) acute fluid overload (AFO) or cardiovascular (CV)-related events. The clinical feasibility of the BCM-BIS algorithm was also inspected. Statistical methods: a software (SAS) 9.3 was used for statistical analysis in this study. R 3.0 was used for graphic presentation of parts of the results. Relative risk, incidence rate ratio and Fisher's exact test were used to compare the discrete outcomes in both groups. Survival analysis was used for time-related events. Repeated-measured and longitudinal data were analyzed with the generalized linear mixed model (GLMM) through the procedure for continuous variables (PROC MIXED) and for discrete variables (PROC GLIMMIX) in SAS.

ELIGIBILITY:
Inclusion Criteria:

MHD patients with age ≥ 18 and dialysis vintage ≥ 3 months

Exclusion Criteria:

1. coronary stents or pacemaker implantation
2. metallic devices in body, such as artificial joints or pins
3. contralateral or bilateral amputations
4. pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 148 | 150
Completed | 128 | 123
Not Completed | 20 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 148 | 150 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (12.1) | 62.1 (11.5) | 62.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 70 | 153
  Male | 65 | 80 | 145

OUTCOME MEASURES:

1. Primary Outcome: All-cause Hospitalization
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: hospitalizations per patient-year
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 128 | 123
hospitalizations per patient-year | 0.52 [0.44 to 0.61] | 0.54 [0.46 to 0.63]

2. Secondary Outcome: Complications During DW Adjustment
Description: we wanted to compared whether the dialysis-related complications are different when DW (dry weight) is adjusted, no matter according to BCM (body composition monitor) results or clinical judgement, in both groups. The result is expressed as the percentage of months in which complications happened when DW adjustment presented (using total months which DW adjustments are present as denominator).
Time Frame: 1 year
Measure: Number; unit: % of months in which compli
Units Other Than Participants: months when dry weight adjustment happen
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 128 | 123
Number analyzed (months when dry weight adjustment happen) | 816 | 735
% of months in which compli | 11.76 | 30.88

ADVERSE EVENTS:
Arm/Group | Study Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/128 | 0/123
Other Adverse Events (participants affected / at risk) | 0/128 | 0/123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes